CLINICAL TRIAL: NCT06037603
Title: Home-based and Mobile App-guided Dual-Task Exercise for Cognition and Functional Capacity After Mild Traumatic Brain Injury (mTBI)
Brief Title: Dual-Task Exercise for Mild Traumatic Brain Injury (mTBI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UNLV-2023-245
Record Dates: First submitted 2023-07-07; First posted 2023-09-14 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-05

CONDITIONS: TBI (Traumatic Brain Injury); Brain Concussion; Clinical Trial; Rehabilitation; Cognition; Psychosocial Functioning; Walking; Vision, Ocular; Mobile Application; Saliva; microRNA; Exercise
Keywords: dual-task exercise; mobile app-guided; home-based; mild traumatic brain injury (mTBI); cognitive function; physical function; psychosocial function; salivary exosomal microRNA
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Concussion; Motor Activity

STUDY DESIGN:
Intervention Model Description: Non-blinded randomized trial with a wait-list control design
Masking Description: Non-blinded randomized trial with a wait-list control design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): The intervention group will be asked to visit the UNLV study site three times to evaluate baseline (T1), post-intervention (T2), and at 1-month post-intervention (T3) for functional assessments and saliva collection. Each participant will complete the BraW-Day program between baseline (T1) and post-intervention (T2). The program consists of 15-minute-long daily cognitive-walking tasks for 14 consecutive days. The program will be delivered on the Uplode mobile app. Each participant will be asked to perform three different 5-minute-long cognitive tasks (e.g., subtracting numbers or remembering long phrases) and one physical task (tandem walking or 8-shape walking) either indoors or outdoors at the same time for 15 minutes every day, which they will repeat daily for the next 13 days (2 weeks in total).
  Interventions: Behavioral: Brain & Walk Exercise Every Day (BraW-Day)
- Wait-list Control (Active Comparator): The wait-list control group will be will be asked to visit the UNLV study site four times to evaluate pre-baseline (T0), baseline (T1), post-intervention (T2), and at 1-month post-intervention (T3) for functional assessments and saliva collection. Each participant will complete the BraW-Day program between baseline (T1) and post-intervention (T2). The program consists of 15-minute-long daily cognitive-walking tasks for 14 consecutive days. The program will be delivered on the Uplode mobile app. Each participant will be asked to perform three different 5-minute-long cognitive tasks (e.g., subtracting numbers or remembering long phrases) and one physical task (tandem walking or 8-shape walking) either indoors or outdoors at the same time for 15 minutes every day, which they will repeat daily for the next 13 days (2 weeks in total).
  Interventions: Behavioral: Brain & Walk Exercise Every Day (BraW-Day)

INTERVENTIONS:
Behavioral: Brain & Walk Exercise Every Day (BraW-Day) — The Brain & Walk Exercise Every Day (BraW-Day) program comprises 15-minute-long daily cognitive-walking tasks for 14 consecutive days. The program will be delivered on the Uplode mobile app. Each participant will be asked to perform three different 5-minute-long cognitive tasks (e.g., subtracting numbers or remembering long phrases) and one physical task (tandem walking or 8-shape walking) either indoors or outdoors at the same time for 15 minutes every day, which they will repeat daily for the next 13 days (2 weeks in total).

SUMMARY:
The investigators previously developed a virtual 14-day dual-task walking exercise program and tested its feasibility with individuals with mild traumatic brain injury (mTBI) history. The investigators will test the feasibility and efficacy of a mobile app-version (Uplode) of the same 14-day exercise program (Brain & Walk Exercise Every Day [BraW-Day]), on cognition, sensorimotor, and other functions in a group of voluntary young adults with an mTBI between last three months to two years, including student athletes, Veterans, and ethnic minorities.

DETAILED DESCRIPTION:
There is a critical need to develop an effective intervention for a chronic concussion or mild traumatic brain injury (mTBI) that presents persistent post-injury functional declines. Up to 40% of mTBIs cause multifaceted and long-term functional declines, including cognitive declines, psychosocial or sensorimotor problems, which results in $17B medical costs each year. Long-term functional impairments have been reported even 5 to 19 years post-injury, which exacerbate neurodegeneration, such as chronic traumatic encephalopathy or Parkinson's disease. Yet, only a very limited or few studies have investigated a followup screening or intervention for long-term and persistent functional declines, suggesting important deficiencies in long-term care for mTBI. The investigators previously developed a virtual 14-day dual-task walking exercise program and tested its feasibility with Asian and Pacific Islanders (API), including those with mTBI history. The investigators will test the feasibility and efficacy of a mobile app-version (Uplode) of the same 14-day exercise program (Brain & Walk Exercise Every Day [BraW-Day]), on cognition, sensorimotor, and other functions in a group of voluntary young adults with an mTBI between last three months to two years, including student athletes, Veterans, and ethnic minorities. The specific aims of the current study are:

Aim 1: Examine if the mobile app, home-based BraW-Day program is acceptable to young adults with an mTBI. H1. BraW-Day program will (a) be acceptable to the participants, (b) fit with their daily life, and (c) demonstrate feasible and suitable data collection of the daily participation.

Aim 2: Test the efficacy of the BraW-Day program on functions after mTBI. H2. BraW-Day program will improve (a) cognitive (measured by a computerized CNS-VS), (b) psychosocial (by Neuro QoL, a standardized self-report tool for neuro-psychosocial conditions), or (c) sensorimotor functions (by walking movement measuring app, 3D kinematic and kinetic gait analysis, and EyeLink rapid eye movement tracker) in mTBI at post-intervention (T2), compared to wait-list controls.

Aim 3: Examine the sustained effect of the BraW-Day program on function after mTBI. H3. Functional levels one month after intervention (T3) will be equivalent to or higher than baseline (T1) and postintervention (T2) levels.

We will conduct a nonblinded randomized trial with a wait-list control design to test the efficacy of a 2-week (14 consecutive days) BraW-Day, which is daily home-based mobile app-based cognitive-walking exercise program on overall functions in individuals with a recent history of mTBI. Both male and female voluntary young adults aged 18 to 40 years with diverse ethnic backgrounds who report a recent history of mTBI, including student athletes and Veterans, will be invited to our exercise intervention. The participants will be randomly assigned to either the intervention group or the control group. Intervention group will have a 3 study visits to ULNV for assessing the baseline (T1), post-intervention (T2), and 1-month post-intervention (T3) functional levels to test the efficacy of the program. The waitlist control group will have an additional study visit at pre-baseline (T0), so will have a total of 4 study visits (T0, T1, T2, & T3). The BraW-Day intervention program consists of 15-minute-long daily brain exercise and walking at the same time (i.e., cognitive-walking tasks) for 14 consecutive days, targeting persistent mTBI symptoms and functional declines, including cognitive, psychosocial, and sensorimotor functions. The BraW Day program will be delivered on a mobile app, Uplode. All subjects will be introduced to the BraW-Day program and the Uplode app. They will be guided to download the Uplode app on their mobile phone with the app's notification enabled for the next day when they will start the BraW-Day program as Day 1. From Day 1, daily reminder notifications from the app will be sent to each participant's mobile phone. They will then follow the schedule for the daily exercise as guided by the app. Each participant will be asked to perform three different 5-minute-long cognitive tasks (e.g., subtracting numbers or remembering long phrases) and one physical task (i.e., tandem walking or 8-shape walking) either indoor or outdoor at the same time for 15 minutes every day, which they will repeat daily for the next 13 days (2 weeks in total). Participants will be asked to mark the start time and the end time of the 15-minute dual-task exercise every day and also to mark off each of the 3 different cognitive tasks every time they finish on that day. Once each participant hits the "Submit" button when they complete each 15-minute-long exercise every day. Post-injury functional levels will be measured by the Rivermead Post-concussion Symptom Questionnaire (RPQ) and the Neurobehavioral symptom inventory (NSI). At each site visit, participants will complete functional assessments (cognitive, psychosocial, sensorimotor function) and collect a saliva sample, which will take est. 1.5 hours per visit. More specifically, cognitive functional assessment will be by a computerized CNS-VS, psychosocial by Neuro QoL (a standardized self-report tool for neuro-psychosocial conditions), and sensorimotor by the mHealth-WB app, 3D kinematic and kinetic gait analysis, and EyeLink rapid eye movement tracker. T2 visit will include a semi-structured interview (max. 20 mins) based on components of the System Usability Scale (SUS) focusing on acceptability, feasibility, and barriers and facilitators for the BraW-Day exercise program on the Uplode app. Saliva samples will be collected and saved for future profiling of peripheral epigenetic markers (i.e., saliva exosomal microRNA). This will be explained as part of informed consent process.

No adverse events are expected from the implementation of the project, including the BraW-Day home-based exercise intervention, based on our previous virtual format of the same intervention. All healthcare providers in the proposed project are board-certified and credentialed in each of their states. All participants will be strongly encouraged to contact and report any adverse event during the study participation. The PI's contact information and a list of campus resources, primary care, and urgent care settings will be shared with every participant in their first site visit. If any adverse events happen during the project, within 24 hours of the discovery of the occurrence, the PI will submit adverse event reports to the UNLV IRB and the CTR-IN Pilot Program committee.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged 18-40 years
* reporting a recent history of mTBI (3 months - 2 years) based on the Ohio State University TBI Identification Method (OSU TBI-ID)
* understanding the protocol, and
* capable of participating in the full BraW-Day program and completing assessments

Exclusion Criteria:

* Those with other active medical disease or such history
* psychiatric disturbance, substance abuse, learning disorder, or attention deficit hyperactivity disorder (ADHD)
* any impairments that may prevent the participant from completing the tests safely, or
* currently on prescribed medications
* involved in any type of legal action related to the mTBI

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-03-06 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Change in cognitive function from baseline at 15 days (Post-intervention) and 45 days (1-month post-intervention) | 45 days
  The CNS-Vital Signs Test is a computerized test of cognitive functioning with good-to-excellent reliabilities (most r's > 0.8) in its different sub-tests. It will measure comprehensive neurocognitive function, including memory, attention psychomotor speed, reaction time, and cognitive flexibility. Higher scores mean better cognitive functioning outcomes. The CNS-Vital Signs Test standard scores and percentile ranks are auto-scored using an algorithm based on a normative data set of 1600+ subjects, ranging from Ages 8 - 90. Standard scores > 110 or percentile scores > 74 indicate high function and high capacity, and standard scores < 70 or percentile scores < 2 indicate deficit and impairment likely.
Change in psychosocial function from baseline at 15 days (Post-intervention) and 45 days (1-month post-intervention) | 45 days
  The Quality of Life in Neurological Disorders Item Bank will be used to assess depressive, anxious symptoms, fatigue, sleep disturbances, and other functions that may be affected by chronic mTBI. Each domain measure has undergone rigorous qualitative and psychometric evaluation and refinement through numerous clinical studies, so the measures could provide efficient, precise, valid, and responsive indicators of a person's health status. Higher scores mean better psychosocial functioning outcomes. The Quality of Life in Neurological Disorders Item Bank scores have a mean of 50 and standard deviation (SD) of 10 in a referent population.
  Scores 0.5 - 1.0 SD worse than the mean = mild symptoms/impairment Scores 1.0 - 2.0 SD worse than the mean = moderate symptoms/impairment Scores 2.0 SD or more worse than the mean = severe symptoms/impairment
Change in sensorimotor function - vision from baseline at 15 days (Post-intervention) and 45 days (1-month post-intervention) | 45 days
  Rapid eye movement by EyeLink 1000 Plus System (SR Research)
Change in sensorimotor function - walking from baseline at 15 days (Post-intervention) and 45 days (1-month post-intervention) | 45 days
  Walking features and balance by mobile health application for walking balance (mHealth-WB)
Change in sensorimotor function - gait from baseline at 15 days (Post-intervention) and 45 days (1-month post-intervention) | 45 days
  3-dimensional kinematic and kinetic gait analysis (lab-based approach)
Acceptability, feasibility of the BraW-Day program on Uplode app | 15 days
  Semi-structured interview (max. 20 mins) based on components of the System Usability Scale focusing on acceptability, feasibility, and barriers and facilitators for the BraW-Day exercise program on the Uplode app. System Usability Scale scores are standardized on a 0-100 scale, Higher scores mean better acceptability of an app, so in this study, the Uplode app.

SECONDARY OUTCOMES:
Change in salivary exosomal microRNA from baseline at 15 days (Post-intervention) and 45 days (1-month post-intervention) | 45 days
  Saliva samples will be collected for future characterization of exosomal microRNAs as potential neurodegenerative biomarkers associated with functional level alterations. This will be explained as part of the informed consent process.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nevada, Las Vegas, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: Undecided